CLINICAL TRIAL: NCT06033027
Title: Influence of Assistive Soft-robotic Glove Use on Actual Arm Use in Daily Life
Brief Title: Arm Use With Soft-robotic Glove
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roessingh Research and Development (Other)
Collaborators: Eurostars (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 85214
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Trauma Injury of Hand Multiple; Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Single case experimental design with multiple baselines
Masking Description: Masking is not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline phase (No Intervention)
- Soft-robotic glove phase (Experimental)
  Interventions: Device: Carbonhand
- Retention phase (No Intervention)

INTERVENTIONS:
Device: Carbonhand — During this phase, participants use the Carbonhand soft-robotic glove system in daily life for 6 weeks to support the performance of daily activities with their affected hand in the home environment. The participants are free to choose for which activities, when and for how long they use the Carbonhand. However, it is recommended to use the Carbonhand at least 180 minutes a week during the most common ADL, such as household activities, dressing/undressing, eating/drinking/cooking, and/or leisure activities.
  Arms: Soft-robotic glove phase

SUMMARY:
This study, aimed at investigating the impact of using a supportive soft-robotic glove on actual arm and hand use in daily life, is designed as a single-case experimental design study. 3-5 patients with limitations in hand function due to trauma-related or neurological conditions are asked to participate. Participants will be asked to use a soft-robotic glove at home for six weeks during daily activities relevant to them, while that glove supports the grip of their most affected hand. For several weeks before, during and after the use of the soft-robotic glove, participants will be asked to do some short tests (wearing an activity meter on both wrists during the day, performing a hand squeeze test under the supervision of the researcher via video call) and to answer some questions related to perceived hand function and well-being (a total of at least 15 times during 12-14 weeks). The present study is a follow-up to previous studies that investigated the effect of (previous versions of) the same robotic glove (Carbonhand; Bioservo Technolo-gies AB, Kista, Sweden) on hand function, in order to better understand and explain the observed therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Experience difficulties in performing ADL due to hand function limitations as a result of trauma-related injury or neurologic disorder
* Being in a chronic/stable phase of disease as judged by their physician
* Able to activate the soft-robotic glove by generating pressure on finger/palm sensors when grasping an object
* Ability to relax an active grip
* Sufficient cognitive status to understand two-step instructions
* Having (corrected to) normal vision
* Able to provide written informed consent
* Living independently

Exclusion Criteria:

* Severe sensory problems of the most-affected hand
* Severe acute pain of the most-affected hand
* Wounds on the hands that can provide a problem when using the glove
* Severe contractures limiting passive range of motion to the extent that the glove can't be donned/activated comfortably
* Co-morbidities limiting functional use/performance of the arms and/or hands
* Severe spasticity of the hand (≥2 points on Ashworth Scale)
* Severe proximal weakness (MRC shoulder elevation<4)
* Used the Carbonhand system in the past 3 months
* Participation in other studies that can affect functional performance of the arm/hand
* Receiving arm-/hand function therapy during the course of the study
* Insufficient digital literacy to conduct video calls
* Insufficient knowledge of the Dutch or English language to understand the purpose or methods of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Actual arm activity | During home assessments: 15 times scheduled intermittently across 12-14 weeks (5x in each of the three study phases), while wearing the MotionWatch for a day during waking hours (ca. 12h).
  The main study parameter is actual arm use as measured by two MotionWatch8 devices, containing an accelerometer, one around each wrist. In essence, the 'raw' accelerometer signal will be transformed into an 'activity count signal'. Actual amount of arm-hand use will then be calculated in several ways, focusing on the duration of use and the intensity of use of the affected arm-hand.

SECONDARY OUTCOMES:
Grip strength | During home assessments: 15 times scheduled intermittently across 12-14 weeks (5x in each of the three study phases), with supervision by researcher on videocall
  The maximal handgrip strength will be measured with a Jamar dynamometer (Patterson medical, Warrenville, IL, USA), in accordance with American Society of Hand Therapist guidelines. Each participant is sitting comfortably with the elbow of the affected arm close to their body, flexed 90 degrees, holding the dynamometer in the affected hand. The other parts of the body is not allowed to move or help to give more strength. The participant has to squeeze the handgrip of the dynamometer maximally for 5 seconds. There will be three attempts and between the different attempts are at least 60 seconds rest. The best of the three attempts will count.
Michigan Hand Outcomes Questionnaire - Question 2 (MHQ-Q2) | During home assessments: 15 times scheduled intermittently across 12-14 weeks (5x in each of the three study phases)
  The original MHQ (total of 57 items) asks a patient's opinion about his hands and his health. This list is used to find out how the patient feels and to what extent he is capable of carrying out daily activities. The problem is mapped out within 6 domains: total hand function, ADL, work situation, work performance, pain, aesthetics and satisfaction. For repeated home assessment, we only ask question 2 A/B (most affected right or left hand) and 2 C (bimanual activities) of the domain ADL. This item consists of a total of 12 statements to rate on a 5-points Likert scale. The scores are normalized afterwards to a range of 0 to 100.
Positive Health questionnaire | During home assessments: 15 times scheduled intermittently across 12-14 weeks (5x in each of the three study phases)
  Huber et al. studied how people think about health. They concluded that the concept of health no longer fits within the definition of the World Health Organization (health as complete wellbeing and absence of disease). The Institute for Positive Health created a tool to gain insight into the positive health of a person. This tool consists of 6 dimensions: bodily functions, mental wellbeing, meaningfulness, quality of life, participation, and daily functioning. Participants complete the questionnaire, resulting in a score between 0 and 10 for each dimension [19]. In our study, an adapted version will be used. Instead of completing a questionnaire consisting of 42 questions, the participants score each of the six dimensions from 0 to 10, as reported by van Velsen et al.
Glove use data | Continuously and automatically during soft-robotic glove use phase (6 weeks) when soft-robotic glove is turned on and activated.
  During the intervention phase, glove use time will be automatically recorded in the Carbonhand system, representing objective, cumulative duration of glove activation (recording is stopped after 2 min of inactivity).
Diary | Continuously during soft-robotic glove use phase (6 weeks) when soft-robotic glove is used
  Diary for subjective reports on amount of use and type of activities performed with affected hand with glove, during the six weeks of glove use.
Motor Activity Log (MAL) | Thee times across 12-14 weeks during evaluations at the end of each study phase (between week 2-4, week 8-10, week 12-14, with exact scheduling depending on randomized length of baseline phase)
  The MAL is a semi-structured questionnaire to explore the self-perceived amount of use (AOU) and quality of movement (QOM) of the affected arm and hand by stroke patients during ADL. This questionnaire consists of 26 activities and has excellent test-retest reliability for both scores of each activity. Each activity is rated by the participant for quality of movement and amount of use of the upper extremity. The possible scores for both aspects ranges from 0 to 5.
Jebsen-Taylor hand function test (JTHFT) | Thee times across 12-14 weeks during evaluations at the end of each study phase (between week 2-4, week 8-10, week 12-14, with exact scheduling depending on randomized length of baseline phase)
  The JTHFT is a reliable and valid test to evaluate functional hand motor function in different patient groups and healthy people of various ages. The test consists of 7 different unilateral hand skill tasks related to ADL: (1) writing a sentence of 24 characters, (2) turning over 7.6- x 12.7-cm cards, (3) picking up small, common objects (e.g., paper clips, coins and bottle caps) and move these to a box, (4) stacking checkers (test of eye-hand coordination), (5) simulated feeding (e.g. teaspoon with beans), (6) picking up large empty cans and (7) moving weighted (450 g) cans. The time of each different task will be recorded in seconds and the different times summed is the total score for the test.
Numerical Pain Rating Scale (NPRS) | Thee times across 12-14 weeks during evaluations at the end of each study phase (between week 2-4, week 8-10, week 12-14, with exact scheduling depending on randomized length of baseline phase)
  The NPRS measures the subjective intensity of pain. The NPRS is an 11-point scale from 0-10: '0'= no pain, '10'= the most intense pain imaginable. Patients select a value that is most in line with the intensity of pain that they have experienced in the last 24 hours. The NPRS has good sensitivity, while producing data that can be statistically analysed.
Michigan Hand Outcome Questionnaire - Dutch Language Version (MHQ-DLV) | Thee times across 12-14 weeks during evaluations at the end of each study phase (between week 2-4, week 8-10, week 12-14, with exact scheduling depending on randomized length of baseline phase)
  The full MHQ-DLV with a total of 57 items [17,18] is administered as questionnaire during each lab visit (pre, post and follow-up). It asks a patient's opinion about his hands and his health. This list is used to find out how the patient feels and to what extent he is capable of carrying out daily activities. The problem is mapped out within 6 domains: total hand function, ADL, work situation, work performance, pain, aesthetics and satisfaction.
Euroqol-5D (EQ-5D) | Thee times across 12-14 weeks during evaluations at the end of each study phase (between week 2-4, week 8-10, week 12-14, with exact scheduling depending on randomized length of baseline phase)
  The EQ-5D generic health index is a standardized instrument that is applicable to a wide range of health conditions and treatments. The first part records self-reported problems on the domains mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is divided into five levels of severity corresponding to no problems, slight problems, moderate problems, severe problems and extreme problems. The second part comprises a visual analogue scale (VAS), described as a "feeling thermometer" rated from 0 (worst imaginable health state) to 100 (best imaginable health state).The EQ-5D is designed for self-completion by respondents. In the present study, the EQ-5D will be used to calculate a preference-based summary index based on TTO techniques in which the value 0 represents death and 1 represents perfect health.
Short-Form (SF-36) | Thee times across 12-14 weeks during evaluations at the end of each study phase (between week 2-4, week 8-10, week 12-14, with exact scheduling depending on randomized length of baseline phase)
  The SF-36 is a 36-item questionnaire to assess health perception of people. It is a well-validated and reliable assessment for measuring health perception. The questionnaire consists of multi-item dimensions about physical and mental well-being of the participant. The scores for all dimensions will be calculated and also the physical and mental component summary scores will be calculated, referred to as PCS-36 (average score of the domains physical functioning, physical role functioning, bodily pain and general health) and MCS-36 (average score of the domains vitality, emotional role functioning, social functioning and mental health), respectively. The scores of the questionnaire will be converted to a 0-100 scale, where a higher score indicates a better quality of life.
Semi-structured interview | One time across 12-14 weeks during evaluation at the end of the intervention phase (between week 8-10, with exact scheduling depending on randomized length of baseline phase)
  A qualitative interview with open-ended questions to get a more thorough understanding about the experience of the participants of using the Carbonhand system during ADL at home and the user-friendliness of the system, will be administered after the glove use period (so only during the post assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Gerdienke Prange, PhD, Principal Investigator — Roessingh Research and Development
Locations (1):
- Roessingh Research and Development, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No